CLINICAL TRIAL: NCT05139849
Title: VAsopressin and STeroids in Addition to Adrenaline in Cardiac Arrest - a Randomized Clinical Trial
Acronym: VAST-A
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tiohundra AB (Industry)
Collaborators: Sahlgrenska University Hospital (Other); Stockholm South General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VAST-A.Studyprotocol.Version_4
Record Dates: First submitted 2021-11-17; First posted 2021-12-01 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2021-11

CONDITIONS: Cardiac Arrest;In-hospital Cardiac Arrest; Methylprednisolone; Vasopressin; Adrenaline; Randomized Clinical Trial
MeSH Terms: conditions — Diabetes Insipidus | interventions — Vasopressins; Methylprednisolone; Hydrocortisone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): Adrenaline, vasopressin and steroids arm (intervention)
  1. At randomization
     1 ml of vasopressin 20 IU/ml will be administered as soon as possible after adrenaline during the five first cycles of drug administration during CPR.
     1 ml metylprednisolone sodium succinate 40 mg/ml will be administered only during the first cycle of drug administration during CPR
  2. In the ICU Hydrocortisone 3 mg/ml At 4 hours post ROSC, and then once daily, surviving patients with post-resuscitation shock will receive an infusion of 100 ml (300 mg hydrocortisone/ d) for ≤ 7 days. From day 8 post ROSC or when vasopressors are not needed the hydrocortisone dos will be reduced daily to 67 ml (200 mg) and 33 ml (100 mg) and then discontinued). Patients with evidence of acute myocardial infarction will receive an infusion of 100 ml (300mg hydrocortisone/ d) for maximum 3 days to prevent retardation of infarct healing.
  Interventions: Drug: Vasopressin; Methylprednisolone; Hydrocortisone
- Control (Placebo Comparator): Adrenaline alone arm (control)
  1. At randomization 1 ml sodium chloride 9 mg/ml (placebo) will be administered as soon as possible after adrenaline during the first five cycle of drug administration during CPR 1 ml sodium chloride 9 mg/ml (placebo) will be administered only during the first cycle of drug administration during CPR
  b In the ICU sodium chloride 9 mg/ml (placebo) At 4 hours post ROSC, and then once daily, surviving patients with post-resuscitation shock will receive an infusion of 100 ml for ≤ 7 days. From day 8 post ROSC or when vasopressors are not needed the dos will be reduced daily to 67 ml and 33 ml and then discontinued. Patients with evidence of acute myocardial infarction will receive an infusion of 100 ml for 3 days.
  Interventions: Drug: Sodium chloride

INTERVENTIONS:
Drug: Vasopressin; Methylprednisolone; Hydrocortisone — Vasopressin, the vasoconstrictive hypophysal hormone, alone has not shown increased survival when compared to adrenaline. However, animal data have shown increased diastolic pressure, cerebral perfusion pressure and cerebral oxygenation in cardiac arrest treatment with vasopressin, and have when compared to adrenaline been associated with better cerebral blood flow.
  Corticosteroids are currently used in septic shock treatment as a means to reduce time to shock reversal and thereby potentially improving mortality. Steroids have therefore also been suggested for cardiac arrest treatment. The potential role in resuscitation includes the catecholaminerg potentiation, vasoconstriction and protection from reperfusion injury.
  Arms: Intervention
Drug: Sodium chloride — Sodium chloride 9 mg/ml
  Arms: Control

SUMMARY:
This is an investigator initiated randomized, placebo controlled, double blind, superiority, multi-centre clinical trial. The estimated study project period runs over 3-4 years, including pilot phase. Based on preliminary assumptions, to confirm or reject an increase in survival from 9% to 14%, about1400 patients will be randomized in the study. In hospital cardiac arrest patients meeting criteria(s) for adrenaline administration according to current ERC guidelines are eligible for randomization in the study.

Informed consent for participating in the study cannot be obtained from the subject at the scene of the cardiac arrest since the victim is unconscious. Therefore, all hospitalized men > 18 years and women > 50 years, except those fulfilling the exclusion criterias; patients not capable to comprehend information to decide about participation in the study, women considered of childbearing potential (WOCBP)) and do not resuscitate (DNR) decision will be informed and asked about consent to participate in the study and in the case of cardiac arrest during the actual hospital stay randomized to either treatment. Only those patients experiencing an in hospital cardiac arrest meeting criteria(s) for adrenaline administration will be randomized.

Patients will be randomized to, in addition adrenaline, either treatment with vasopressin and steroids (intervention) or sodium chloride (placebo) (control).

Primary outcome is survival at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized men > 18 years and hospitalized women > 50 years.

Exclusion Criteria:

* Patients not capable to comprehend information to decide about participation in the study
* Women considered of childbearing potential (WOCBP) i. e. premenopausal women
* Patients with do not resuscitate (DNR) descision
* Prior enrollment and randomization in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1276 (Estimated)
Dates: Start 2021-11-17 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Survival at 30 days | Survival at 30 days
  Survival at 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Sune Forsberg, MD, PhD, Principal Investigator — Tiohundra AB; Peter Lundgren, MD, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (2):
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Tiohundra, Norrtälje

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andersen LW, Holmberg MJ, Hoybye M, Isbye D, Kjaergaard J, Darling S, Zwisler ST, Larsen JM, Rasmussen BS, Iversen K, Schultz M, Sindberg B, Fink Valentin M, Granfeldt A. Vasopressin and methylprednisolone and hemodynamics after in-hospital cardiac arrest - A post hoc analysis of the VAM-IHCA trial. Resuscitation. 2023 Oct;191:109922. doi: 10.1016/j.resuscitation.2023.109922. Epub 2023 Aug 3. PMID 37543161